CLINICAL TRIAL: NCT04721145
Title: IMPaCT: IMPlementing Continuous Glucose Monitoring in High-risk, Poorly Controlled Children With Type 1 Diabetes
Brief Title: CGM Use in Poorly Controlled Youth With Type 1 Diabetes
Acronym: IMPaCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00255470
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes; Hypoglycemia; High Blood Sugar
Keywords: Continuous Glucose Monitoring; Time in range; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dexcom G6 Continuous Glucose Monitor (Experimental): Children with type 1 diabetes will wear a continuous glucose monitor (CGM) for 10 days.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitor

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitor — Eligible patients will have a Dexcom G6 Continuous Glucose Monitor placed for 10 days.

SUMMARY:
The purpose of this prospective study is to determine if trial use of a Dexcom G6 CGM system for a 10 day wear period in high risk, poorly controlled pediatric Type 1 diabetes patients increases uptake of personal CGM use, and improves short-term time in range glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 diabetes for >3 months

Exclusion Criteria:

* CGM use in the last 6 months

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa Wolf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Pediatric Diabetes Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phu A, Lin T, Manfredo JA, Brown EA, Wolf RM. Similar Perceptions on Continuous Glucose Monitor Use amongst Youth with Type 1 and Type 2 Diabetes. Pediatr Diabetes. 2023 Jun 19;2023:1979635. doi: 10.1155/2023/1979635. eCollection 2023. PMID 40303266
- [Derived] Lin T, Manfredo JA, Illesca N, Abiola K, Hwang N, Salsberg S, Akhtar Y, Mathioudakis N, Brown EA, Wolf RM. Improving Continuous Glucose Monitoring Uptake in Underserved Youth with Type 1 Diabetes: The IMPACT Study. Diabetes Technol Ther. 2023 Jan;25(1):13-19. doi: 10.1089/dia.2022.0347. Epub 2022 Nov 7. PMID 36223197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 11
  Race/Ethnicity: Non-Hispanic Black | 11
  Race/Ethnicity: Hispanic | 3
  Race/Ethnicity: Multi-racial (American Indian / White) | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Insurance [Count of Participants; unit: Participants] — Type of insurance participant was using at time of enrollment, collected from the medical record.
  Participants
    Public Insurance | 17
    Private Insurance | 9
HbA1c [Mean (Standard Deviation); unit: Percentage] | 10.7 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Personal CGM Use
Description: Evaluate whether there is any change in uptake of personal CGM after 10-day trial.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 26
Participants
  Wants a personal CGM | 22
  Does not want a personal CGM | 4

2. Secondary Outcome: Change in the Percent Time in Range Glucose Control
Description: Changes in time in range glucose control from 1-5 days to 6-10 days from the Dexcom CGM
Time Frame: 1-5 days and 6-10 days
Population: Only 15/26 participants had data from both periods
Measure: Mean (Standard Deviation); unit: Percentage of time in range
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 15
Percentage of time in range
  1-5 days | 41.9 (21.2)
  6-10 days | 32.8 (15.2)

3. Secondary Outcome: Change in Hemoglobin A1c
Description: Changes in HbA1c from baseline to next available A1c at 3-6 month follow up visit
Time Frame: Baseline, 3-6 months
Population: 20/26 participants had a follow up A1c lab available.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 20
Percentage
  Baseline | 10.9 (2.6)
  3-6 month follow up | 10.8 (2.6)

4. Secondary Outcome: Using Personal CGM
Description: Percentage of participants using CGM at time of follow up, of those who reported wanting a personal CGM
Time Frame: 3-6 months
Population: 21/26 participants wanted a personal CGM AND completed 3-6 month follow-up. (Of the total participants 4 participants did not want CGM. 1 participant had no 3-6 month follow up. Thus, this analysis includes the remaining 21 participants.)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 21
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dexcom G6 Continuous Glucose Monitor
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 5/26
Other Adverse Events (participants affected / at risk) | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom G6 Continuous Glucose Monitor (N=26)
DKA admission (Endocrine disorders) | 4 (4) — Admission for diabetic ketoacidosis
ER Visit, renal stone (Renal and urinary disorders) | 1 (1) — Kidney Stone
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Hospitalization due to severe abdominal pain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom G6 Continuous Glucose Monitor (N=26)
Otalgia of both ears (Ear and labyrinth disorders) | 1 (1) — Otalgia of both ears, seen in ER, middle ear effusions.

LIMITATIONS AND CAVEATS:
The patient cohort was small, and may not be generalizable to all patients with T1D. Further, the mean HbA1c of individuals in the study was well above ADA target, and the impact of trial CGM on patients with HbA1c closer to goal ADA range may be different. Additionally, follow-up CGM data was not available for most patients, thus limiting data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04721145/Prot_SAP_001.pdf